CLINICAL TRIAL: NCT02606721
Title: An Exploratory Pilot Study Evaluating Various Diagnostic Measurements Taken During an Escalating Dose Oral Food Challenge to Patient Response
Brief Title: Food Allergy Challenge Diagnostic Study
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ORA-FA-001
Record Dates: First submitted 2015-11-10; First posted 2015-11-17 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2016-05

CONDITIONS: Food Hypersensitivity
Keywords: Food Hypersensitivity; Oral Food Challenge; Skin Prick Test; Food Biomarkers
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Challenge Subjects: Male or female subjects aged 5 - 35 with suspected food allergy and an upcoming scheduled clinical food challenge

SUMMARY:
The objective of this study is to correlate various diagnostic measurements taken during an escalating dose oral food challenge to the subject's response. This study will investigate whether non invasive objective biomarkers can indicate a positive response to an escalating dose OFC before a systemic reaction occurs.

DETAILED DESCRIPTION:
Patients often discover their food allergies after consuming a given food and experiencing a subsequent allergic reaction. The majority of patients (75%) will then consult a food allergist for formal diagnosis and treatment information. With respect to patient quality of life, there is tremendous benefit in having a confirmed diagnosis of food allergy as often patients are unsure of the source of their reaction outside the office. Allergists will conduct a Skin Prick Test (SPT) and assess serum specific IgE levels to screen for specific food protein sensitivities. However, a positive response in SPT and specific IgE will confirm only sensitivity, and in more than 70% of cases patients that respond positively to SPT and specific IgE testing will NOT manifest an allergic response to food consumption. To address this issue, most food allergists will recommend an oral food challenge in a controlled setting to confirm the allergic response from consuming the suspected foods. The oral food challenge (OFC) consists of consuming escalating levels of the suspect food, (usually mixed in applesauce or controlled baked goods), until either a reaction manifests or until the challenge is complete with no reaction. The food challenge process poses significant risk to the patient. In 5% of cases, the patient experiences a severe allergic response which requires the use of epinephrine. These responses typically consist of severe reactions in GI or respiratory and arise from challenging patients with higher doses of food allergen then is necessary to prove a mild allergic response, which is directly linked to variability in diagnosis of a positive response, within subjects and within investigators.

The investigators hypothesize that measurements taken using minimally-invasive diagnostic tests during the course of an escalating-dose oral food challenge will be able to detect a positive response before a systemic reaction occurs in the patient and may be able to screen with individuals predisposed to EOE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, aged 5 - 35 years with planned clinical oral food challenge;
* Have provided verbal and written informed consent. If under the age of 18, a parent/guardian must provide verbal and written informed consent;
* Be willing and able to follow instructions, including participation in study assessments, and can be present for the required study visits for the duration of the study;

Exclusion Criteria:

* Be unable to comply with all study parameters and procedures

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with suspected food allergy and scheduled upcoming oral food challenge will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Correlation between objective biomarker measures and challenge outcome | Change from baseline at 15 minute intervals until completion of challenge (approximately 3 hours)
  Correlation between imaging measurements taken before, during, and after oral food challenge to outcome of challenge
Correlation between subjective biomarker measures and challenge outcome | Change from baseline at 15 minute intervals until completion of challenge (approximately 3 hours)
  Correlation between symptom questionnaire taken before, during, and after oral food challenge to outcome of challenge

CONTACTS AND LOCATIONS:
Overall Officials: John Leung, M.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No